CLINICAL TRIAL: NCT02019589
Title: A Phase 3, Randomized, Three-Cycle, Double-Blind, Placebo-Controlled Study to Evaluate Induction of Secretory Conversion of Endometrium and Withdrawal Bleeding After Administration of TX-12-002-HR in Estrogen-Primed Women With Secondary Amenorrhea
Brief Title: A Phase 3, Randomized, Three-Cycle, Double-Blind, Placebo-Controlled Study to Evaluate Induction of Secretory Conversion of Endometrium and Withdrawal Bleeding for Secondary Amenorrhea
Acronym: SPRY
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: TherapeuticsMD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TXP13-01
Record Dates: First submitted 2013-12-18; First posted 2013-12-24 (Estimated); Last update posted 2018-05-08 (Actual); Status verified 2018-05

CONDITIONS: Secondary Amenorrhea
Keywords: Secondary Amenorrhea; SPRY Trial
MeSH Terms: interventions — Progesterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Progesterone 225 mg/day (Active Comparator): Progesterone + Placebo
  Interventions: Drug: Progesterone; Drug: Placebo
- Progesterone, 300 mg/ day (Active Comparator): Progesterone + Placebo
  Interventions: Drug: Progesterone; Drug: Placebo
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Progesterone
  Arms: Progesterone 225 mg/day; Progesterone, 300 mg/ day
Drug: Placebo

SUMMARY:
This study will be a Phase 3, randomized, three-cycle, double-blind, placebo-controlled, parallel group, multiple-dose design.

The study design has four phases: Screening Period; Open-Label Estrogen-Priming Period (Run-In Period); Blinded Treatment Period; and Follow-Up. The Open Label Priming Period and Blinded Treatment Period cover a total of three 28-day cycles. Clinical evaluations will be performed at the following time points:

Screening Period:

• Screening Period (approximately 42 Days)

Open-Label Estrogen Priming Period (Run In Period):

* Visit 1 Baseline (Cycle 1, Day 1)
* Telephone Interview (Cycle 1, Day 28 [- 3 d to ±1d])

Blinded Treatment Period:

* Visit 2 Randomization (Cycle 2, Day 12 [±2d])
* Visit 3 Interim (Cycle 3, Day 12 [±2d])
* Visit 4 End of treatment (Cycle 3, Day 24 [±1d])

Follow-Up Period:

* Visit 5 Follow-Up (Approximately 10 days after the last treatment)
* Telephone Interview (Approximately 2-4 weeks after completion of progestin course) (Only applies to subjects receiving an approved progestin therapy for proliferative endometrium, as determined by biopsy.)

ELIGIBILITY:
Inclusion Criteria:

* Be female, premenopausal, 18 to 40 years of age (inclusive, at the time of randomization)
* Have secondary amenorrhea, defined as the absence of menstruation for at least 90 days prior to Visit 1 (Cycle 1, Day 1).
* Have an intact uterus.
* Be otherwise healthy, as judged by the Investigator physician, based on a medical evaluation performed during the screening period prior to the initial dose of Estrace®. The medical evaluation must include:

  * a normal or non-clinically significant physical examination, including vital signs (sitting blood pressure, heart rate, respiratory rate and temperature). Acceptable sitting systolic blood pressure is <140 mmHg and diastolic blood pressure is <90 mmHg at screening. A subject may be taking up to two antihypertensive medications.
  * a normal or non-clinically significant pelvic examination performed during screening.
  * a normal or non-clinically significant clinical breast examination performed during screening. An acceptable breast examination is defined as no masses, adenopathy, or other findings identified that are suspicious of malignancy.
  * a normal or non-clinically significant 12-lead ECG as determined by the Principal Investigator (PI) or medical Sub-Investigator.
* Have a negative serum pregnancy test at Screening, and be willing to use an acceptable form of non-hormonal birth control (e.g., barrier method with spermicide) during the study. (The "rhythm method," withdrawal, or an IUD are NOT acceptable methods.)

Exclusionary:

* Be postmenopausal.
* Be diagnosed with primary amenorrhea.
* Have had bilateral oophorectomy and/or hysterectomy.
* Have a history of thrombosis of deep veins or arteries or a thromboembolic disorder.
* Have a history of coronary artery or cerebrovascular disease (e.g., myocardial infarction, stroke, TIA).
* Have a history of liver or kidney dysfunction/disorder (e.g., hepatitis C or chronic renal failure).
* Have a history of gallbladder dysfunction/disorders (e.g., cholangitis, cholecystitis), unless gallbladder has been removed.
* Have a history of diabetes, thyroid disease or any other endocrine disease. (Subjects with diet-controlled diabetes or controlled hypothyroid disease at screening are not excluded.)
* Have a history of undiagnosed vaginal bleeding.
* Have any history of endometrial hyperplasia, uterine/endometrial, breast or ovarian cancer.
* Have any history of malignancy within the last 5 years, with the exception of basal cell (excluded if within one year) or squamous cell (excluded if within one year) carcinoma of the skin.
* Have a history of any other cardiovascular, hepatic, renal, pulmonary, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, psychological, or musculoskeletal disease or disorder that is clinically significant in the opinion of the Principal Investigator or medical Sub-Investigator.
* Have used injectable or implantable estrogen, progestin/progesterone, testosterone or androgens within the last 6 months prior to Visit 1 or plan to use them during the study.
* Have used any of the following hormonal products within the last 90 days prior to Visit 1 or plan to use them during the study:

  * Vaginal nonsystemic hormonal products (rings, creams, gels) or vaginal systemic hormonal products (e.g., FemRing).
  * Transdermal estrogen alone or combination estrogen and progestin/progesterone products.
  * Oral hormonal birth control or oral estrogen and/or progestin/progesterone therapy.
  * Percutaneous estrogen lotions/gels.
* Have used oral, topical, vaginal, or patch testosterone or androgen therapy within the last 8 weeks (56 days) prior to Visit 1 or plan to use them during the study.
* Have used injectable corticosteroids within the last 42 days prior to Visit 1 or plan to use them during the study.
* Have used an IUD (either hormonal or non-hormonal) within the previous 90 days prior to Visit 1 or plan to use one during the study.
* Have used, within 28 days prior to the initial dose of Estrace® at Baseline Visit 1, or plan to use during the study, any prescription or over-the-counter (OTC) medications (including herbal products, such as St. John's Wort) that would be expected to alter progesterone activity. (For additional details, see Concomitant and Prohibited Medications, Section 4.3.
* Have participated in another clinical trial within 30 days prior to screening, have received an investigational drug within the 90 days prior to the initial dose of Estrace®, or be likely to participate in a clinical trial or receive another investigational medication during the study.
* Have contraindication to any planned study assessments (e.g., endometrial biopsy).

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2014-01-20 (Actual); Primary Completion 2014-10-31 (Actual); Study Completion 2014-10-31 (Actual)

PRIMARY OUTCOMES:
• The proportion of subjects at Cycle 3 Day 24 ± 1 day on active treatment compared to placebo with complete secretory activity on endometrial biopsy. | 3 Cycles

SECONDARY OUTCOMES:
• The proportion of subjects at Cycle 3 Day 24 ± 1 day on active treatment compared to placebo with total secretory activity (defined as the aggregate of partial and complete secretory activity) on endometrial biopsy. | 3 cycles

CONTACTS AND LOCATIONS:
Locations (22):
- United States (22):
  - Precision Trials/New Horizons Women's Care, Chandler, Arizona
  - Precision Clinical Trials/Arizona Wellness Center for Women, Phoenix, Arizona
  - Visions Clinical Research, Tucson, Arizona
  - California Family Health Council, Berkeley, California
  - California Family Health Council, Los Angeles, California
  - Clinical Research Consulting, Milford, Connecticut
  - Nature Coast Clinical Research, Crystal River, Florida
  - Comprehensive Clinical Trials, LLC, West Palm Beach, Florida
  - Cypress Medical Research Center, Wichita, Kansas
  - Women's Clinic of Lincoln, P.C., Lincoln, Nebraska
  - Lawrence OB-Gyn Clinical Research, Lawrenceville, New Jersey
  - Suffolk OBGYN, Port Jefferson, New York
  - Wake Research Associates, Raleigh, North Carolina
  - Lyndhurst Clinical Research, Winston-Salem, North Carolina
  - University of Cincinnati Physicians Company, Cincinnati, Ohio
  - HWC Women's Research Center, Englewood, Ohio
  - Vista Clinical Research, Columbia, South Carolina
  - Chattanooga Medical Research, Chattanooga, Tennessee
  - Methodist Charlton Medical Center, DeSoto, Texas
  - The Woman's Hospital of Texas Clinical Research Center, Houston, Texas
  - PRO/Salt Lake Women's Center, Sandy City, Utah
  - Tidewater Clinical Research, Virginia Beach, Virginia